CLINICAL TRIAL: NCT05407025
Title: Targeting Inflammation for Endometrial Cancer Prevention
Status: Active, not recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-001880; NCI-2021-14231 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-05-26; First posted 2022-06-07 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen collection): Patients complete a risk factor questionnaire over 15 minutes. Patients also undergo collection of blood and urine during pre-operative visit and collection of tissue samples at the time of surgery.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, urine, and tissue samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Complete risk factor questionnaire

SUMMARY:
This study examines risk assessment and identifies prevention strategies for endometrial cancer. Collecting samples of blood and urine and risk assessments from patients with benign conditions or endometrial cancer may help doctors learn if there is a relationship between chronic inflammation and increase in risk for endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To develop a model for a biobank that can be expanded across the Mayo Enterprise and implemented at extramural collaborative sites, including underserved populations.

OUTLINE: This is an observational study.

Patients complete a risk factor questionnaire over 15 minutes. Patients also undergo collection of blood and urine during pre-operative visit and collection of tissue samples at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 years old undergoing hysterectomy for any benign indication or endometrial cancer

Exclusion Criteria:

* Men
* Women under the age of 18 years
* Women with a history of cancer, except for endometrial cancer or non-melanoma skin cancer
* Women with type 1 diabetes
* Women that have received radiation or chemotherapy for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing hysterectomy at University of North Carolina (UNC) and Mayo Clinic, Florida
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Levels of eicosanoids and specialized pro-resolving mediators (SPMs) in visceral adipose tissue (VAT) | Through study completion, up to 24 weeks
  Will compare eicosanoid and SPM levels by case-control status (women with endometrial carcinoma and women with non-cancerous conditions) in all patients with linear models, adjusted for age and body mass index (BMI) (and menstrual date, if needed).

SECONDARY OUTCOMES:
Ribonucleic acid (RNA) expression pathways related to inflammation in VAT | Through study completion, up to 24 weeks
  Will assess RNA data with cluster analysis and principal component analysis, focusing on inflammatory / immune pathways pathways in 10 patients with endometrioid endometrial cancer and 10 patients with benign conditions, frequency matched on age and body mass index (BMI). We will Will assess RNA expression patterns in relation to eicosanoid / SPMs that discriminate cases versus controls.

CONTACTS AND LOCATIONS:
Overall Officials: Mark E. Sherman, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials